CLINICAL TRIAL: NCT04331912
Title: Outcomes of Patients With Advanced Neuroendocrine Cancer (NEN) Treated With Systemic Treatment: Somatostatin Analogues, Molecular Targeted Therapy, Chemotherapy and Peptide Radioisotope Therapy - a Retrospective Analysis.
Brief Title: PFS and OS of Patients With Advanced Neuroendocrine Cancer (NEN) After Systemic Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Warmia and Mazury (Other)
Responsible Party: Principal Investigator, Jaroslaw B. Cwikla, MD, PhD, Professor UWM, MD, PhD, Professor UWM, University of Warmia and Mazury
Other Study IDs: NEN_2019
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Neuroendocrine Tumors
Keywords: NEN-neuroendocrine cancer, overall survival; OS - overall survival; PFS - progression-free survival
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study. The analysis includes patients with advanced neuroendocrine cancer (NEN) treated with systemic therapy, because of inoperable primary tumor or/and metastasis, clinical, imaging, biochemical disease progression and no standard method of treatment hormone overproduction symptoms. The data of patients with advanced NEN with histopathological confirmation is collected from medical records. The progression-free survival (PFS), overall survival (OS) and influence of various factors on survival will be estimated. The research will be conducted for above 3 years on planned group 1500 patients. The aim of the study is to estimate median OS and PFS in advanced NEN patients treated with different schedule of systemic treatment.

DETAILED DESCRIPTION:
This is a retrospective study. The analysis includes patients with advanced neuroendocrine cancer (NEN) treated with systemic therapy, because of inoperable primary tumor or/and metastasis, clinical, imaging, biochemical disease progression and no standard method of treatment hormone overproduction symptoms. Systemic treatment including: somatostatin receptor analogues, molecular targeted therapy (sunitinib and everolimus), chemotherapy and peptide radioisotope therapy (Peptide Receptor Radionuclide Therapy). The data of patients with advanced NEN with histopathological or/and clinical or/and biochemical confirmation is collected from medical records. Neuroendocrine cancer from digestive system, respiratory system and another rarely occurring cancer including cancer connected with genetic syndromes like: MEN1, MEN2, VHL, NF1, SDHx will be included. The progression-free survival (PFS), overall survival (OS) and influence of various factors on survival will be estimated. Analyzed factors: age, sex, ethnicity, specific symptoms at the time of diagnosis, carcinoid heart disease, level of 5HIAA in DZM, level of CgA, liver test, size of tumor, cell differentiation of tumor based on Ki-67 index, liver metastases. The research will be conducted for above 3 years since July 2019 till December 2022 on planned group 1500 patients. The aim of the study is to estimate median OS and PFS in advanced NEN patients treated with different schedule of systemic treatment. The second goal is to create clinical practice recommendation based on potential prognostic factors of OS and PFS due to type of therapy in different NEN subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old, male or female,
* Patients with histopathological confirmation of advanced neuroendocrine cancer (NEN),
* Patients with NETG1, NETG2 based on Ki-67,
* Patients with diagnosed NEN, who did not receive prior treatment and were qualified to systemic treatment,
* Patients with advanced NEN who previously received first-line systemic therapy or second-line systemic therapy,
* Patients with advanced, inoperable NEN cancer before the treatment, during the treatment and after the treatment regardless of lines of systemic therapy,
* Patients with diagnosed NEN and performance status (PS) ≤3 according to ECOG/WHO classification, who received systemic therapy.

Exclusion Criteria:

* Patients without histopathological confirmation of neuroendocrine carcinoma (NEN),
* Patients with diagnosed another type of cancer or benign tumor confirmed in histopathological examination,
* Patients treated prior with intention to treat (ITT),
* Patients with residual disease in further clinical follow-up without active systemic treatment,
* Patients with advanced, progressive and poor performance status, who were disqualified from further systemic treatment,
* Patients, who finished treatment during first month or their further disease process was unknown.

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is planned on a group 1500 patients with advanced, histopathologically confirmed neuroendocrine neoplasms (NEN) treated with different schedule of systemic treatment including: somatostatin receptor analogues, molecular targeted therapy (sunitinib or everolimus), chemotherapy using different therapeutic regimens and peptide receptor radioisotope therapy (Peptide Receptor Radionuclide Therapy).
  Research on NEN patients will include the following groups of patients:
  1. NEN from digestive system,
  2. respiratory system;
  3. Other NEN tumours including PPGL, cancer of known primary and very rare NEN tumours like gynecological or urological primary NET.
  4. NEN connected with genetic syndromes like: MEN1, MEN2, VHL, NF1, SDHx.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS - Progression Free Survival | 7 years
  the time from the start of systemic treatment date to the date of first documented disease progression (event: disease progression - DP, based on RECIST, death, adverse events, which provide to disqualification from further therapy). Patients without progression at the time of analysis will be censored.
OS - Overall Survival | 7 years
  is defined as the time from the start of systemic treatment date to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.

SECONDARY OUTCOMES:
Log-rank test | 7 years
  assessment of differences in survival of patients between subgroups
Cox proportional-hazards model | 7 years
  uni- and multivariate analyses used for investigating the association between the survival time of patients and prognostic factors

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - University of Warmia and Mazury in Olsztyn, Olsztyn, Warmian-Masurian Voivodeship
  - Diagnostic and Therapy Center - Gammed, Warsaw

REFERENCES:
- [Result] Modlin IM, Shapiro MD, Kidd M. Siegfried Oberndorfer: origins and perspectives of carcinoid tumors. Hum Pathol. 2004 Dec;35(12):1440-51. doi: 10.1016/j.humpath.2004.09.018. PMID 15619202
- [Result] Modlin IM, Oberg K, Chung DC, Jensen RT, de Herder WW, Thakker RV, Caplin M, Delle Fave G, Kaltsas GA, Krenning EP, Moss SF, Nilsson O, Rindi G, Salazar R, Ruszniewski P, Sundin A. Gastroenteropancreatic neuroendocrine tumours. Lancet Oncol. 2008 Jan;9(1):61-72. doi: 10.1016/S1470-2045(07)70410-2. PMID 18177818
- [Result] Modlin IM, Champaneria MC, Bornschein J, Kidd M. Evolution of the diffuse neuroendocrine system--clear cells and cloudy origins. Neuroendocrinology. 2006;84(2):69-82. doi: 10.1159/000096997. Epub 2006 Nov 9. PMID 17106184
- [Result] Modlin IM, Lye KD, Kidd M. A 5-decade analysis of 13,715 carcinoid tumors. Cancer. 2003 Feb 15;97(4):934-59. doi: 10.1002/cncr.11105. PMID 12569593
- [Result] Kloppel G, Perren A, Heitz PU. The gastroenteropancreatic neuroendocrine cell system and its tumors: the WHO classification. Ann N Y Acad Sci. 2004 Apr;1014:13-27. doi: 10.1196/annals.1294.002. PMID 15153416
- [Result] Greene FL. TNM staging for malignancies of the digestive tract: 2003 changes and beyond. Semin Surg Oncol. 2003;21(1):23-9. doi: 10.1002/ssu.10018. PMID 12923913
- [Result] Kloppel G, Rindi G, Perren A, Komminoth P, Klimstra DS. The ENETS and AJCC/UICC TNM classifications of the neuroendocrine tumors of the gastrointestinal tract and the pancreas: a statement. Virchows Arch. 2010 Jun;456(6):595-7. doi: 10.1007/s00428-010-0924-6. Epub 2010 Apr 27. No abstract available. PMID 20422210
- [Result] Washington MK, Tang LH, Berlin J, Branton PA, Burgart LJ, Carter DK, Compton CC, Fitzgibbons PL, Frankel WL, Jessup JM, Kakar S, Minsky B, Nakhleh RE; Members of the Cancer Committee, College of American Pathologists. Protocol for the examination of specimens from patients with neuroendocrine tumors (carcinoid tumors) of the small intestine and ampulla. Arch Pathol Lab Med. 2010 Feb;134(2):181-6. doi: 10.5858/134.2.181. No abstract available. PMID 20121604
- [Result] Rindi G, Kloppel G, Couvelard A, Komminoth P, Korner M, Lopes JM, McNicol AM, Nilsson O, Perren A, Scarpa A, Scoazec JY, Wiedenmann B. TNM staging of midgut and hindgut (neuro) endocrine tumors: a consensus proposal including a grading system. Virchows Arch. 2007 Oct;451(4):757-62. doi: 10.1007/s00428-007-0452-1. Epub 2007 Aug 3. PMID 17674042
- [Result] Klimstra DS, Modlin IR, Adsay NV, Chetty R, Deshpande V, Gonen M, Jensen RT, Kidd M, Kulke MH, Lloyd RV, Moran C, Moss SF, Oberg K, O'Toole D, Rindi G, Robert ME, Suster S, Tang LH, Tzen CY, Washington MK, Wiedenmann B, Yao J. Pathology reporting of neuroendocrine tumors: application of the Delphic consensus process to the development of a minimum pathology data set. Am J Surg Pathol. 2010 Mar;34(3):300-13. doi: 10.1097/PAS.0b013e3181ce1447. PMID 20118772
- [Result] Modlin IM, Gustafsson BI, Pavel M, Svejda B, Lawrence B, Kidd M. A nomogram to assess small-intestinal neuroendocrine tumor ('carcinoid') survival. Neuroendocrinology. 2010;92(3):143-57. doi: 10.1159/000319784. Epub 2010 Aug 23. PMID 20733279
- [Result] Delle Fave G, O'Toole D, Sundin A, Taal B, Ferolla P, Ramage JK, Ferone D, Ito T, Weber W, Zheng-Pei Z, De Herder WW, Pascher A, Ruszniewski P; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for Gastroduodenal Neuroendocrine Neoplasms. Neuroendocrinology. 2016;103(2):119-24. doi: 10.1159/000443168. Epub 2016 Jan 19. No abstract available. PMID 26784901
- [Result] Niederle B, Pape UF, Costa F, Gross D, Kelestimur F, Knigge U, Oberg K, Pavel M, Perren A, Toumpanakis C, O'Connor J, O'Toole D, Krenning E, Reed N, Kianmanesh R; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for Neuroendocrine Neoplasms of the Jejunum and Ileum. Neuroendocrinology. 2016;103(2):125-38. doi: 10.1159/000443170. Epub 2016 Jan 12. No abstract available. PMID 26758972
- [Result] Ramage JK, De Herder WW, Delle Fave G, Ferolla P, Ferone D, Ito T, Ruszniewski P, Sundin A, Weber W, Zheng-Pei Z, Taal B, Pascher A; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for Colorectal Neuroendocrine Neoplasms. Neuroendocrinology. 2016;103(2):139-43. doi: 10.1159/000443166. Epub 2016 Jan 5. No abstract available. PMID 26730835
- [Result] Pape UF, Niederle B, Costa F, Gross D, Kelestimur F, Kianmanesh R, Knigge U, Oberg K, Pavel M, Perren A, Toumpanakis C, O'Connor J, Krenning E, Reed N, O'Toole D; Vienna Consensus Conference participants. ENETS Consensus Guidelines for Neuroendocrine Neoplasms of the Appendix (Excluding Goblet Cell Carcinomas). Neuroendocrinology. 2016;103(2):144-52. doi: 10.1159/000443165. Epub 2016 Jan 5. No abstract available. PMID 26730583
- [Result] Falconi M, Eriksson B, Kaltsas G, Bartsch DK, Capdevila J, Caplin M, Kos-Kudla B, Kwekkeboom D, Rindi G, Kloppel G, Reed N, Kianmanesh R, Jensen RT; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for the Management of Patients with Functional Pancreatic Neuroendocrine Tumors and Non-Functional Pancreatic Neuroendocrine Tumors. Neuroendocrinology. 2016;103(2):153-71. doi: 10.1159/000443171. Epub 2016 Jan 5. No abstract available. PMID 26742109
- [Result] Pavel M, O'Toole D, Costa F, Capdevila J, Gross D, Kianmanesh R, Krenning E, Knigge U, Salazar R, Pape UF, Oberg K; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for the Management of Distant Metastatic Disease of Intestinal, Pancreatic, Bronchial Neuroendocrine Neoplasms (NEN) and NEN of Unknown Primary Site. Neuroendocrinology. 2016;103(2):172-85. doi: 10.1159/000443167. Epub 2016 Jan 5. No abstract available. PMID 26731013
- [Result] Garcia-Carbonero R, Sorbye H, Baudin E, Raymond E, Wiedenmann B, Niederle B, Sedlackova E, Toumpanakis C, Anlauf M, Cwikla JB, Caplin M, O'Toole D, Perren A; Vienna Consensus Conference participants. ENETS Consensus Guidelines for High-Grade Gastroenteropancreatic Neuroendocrine Tumors and Neuroendocrine Carcinomas. Neuroendocrinology. 2016;103(2):186-94. doi: 10.1159/000443172. Epub 2016 Jan 5. No abstract available. PMID 26731334
- [Result] Peczkowska M, Erlic Z, Hoffmann MM, Furmanek M, Cwikla J, Kubaszek A, Prejbisz A, Szutkowski Z, Kawecki A, Chojnowski K, Lewczuk A, Litwin M, Szyfter W, Walter MA, Sullivan M, Eng C, Januszewicz A, Neumann HP. Impact of screening kindreds for SDHD p.Cys11X as a common mutation associated with paraganglioma syndrome type 1. J Clin Endocrinol Metab. 2008 Dec;93(12):4818-25. doi: 10.1210/jc.2008-1290. Epub 2008 Sep 30. PMID 18826997
- [Result] Iasonos A, Schrag D, Raj GV, Panageas KS. How to build and interpret a nomogram for cancer prognosis. J Clin Oncol. 2008 Mar 10;26(8):1364-70. doi: 10.1200/JCO.2007.12.9791. PMID 18323559